CLINICAL TRIAL: NCT00606645
Title: A Phase 1 Study of Every Other Week XmAb®2513 to Evaluate the Safety, Tolerability, and Pharmacokinetics in Patients With Hodgkin Lymphoma or Anaplastic Large Cell Lymphoma
Brief Title: Safety Study of XmAb®2513 to Treat Hodgkin Lymphoma or Anaplastic Large Cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XmAb2513-01
Record Dates: First submitted 2008-01-21; First posted 2008-02-04 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Hodgkin Lymphoma; Anaplastic Large Cell Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic | interventions — XMAB-2513

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): XmAb2513
  Interventions: Biological: XmAb2513

INTERVENTIONS:
Biological: XmAb2513 — Intravenous infusion of XmAb2513 administered at a dose of 0.3, 1.0, 3.0, 6.0, 9.0, or 12 mg/kg in sequential dose cohorts.

SUMMARY:
An open-label, multi-dose, single-arm, Phase 1 dose escalation study of XmAb®2513 was conducted to define the MTD or recommended dose(s) for further study, to determine safety and tolerability, to characterize PK and immunogenicity, and to evaluate antitumor activity of XmAb2513 in patients with HL and ALCL (non-cutaneous) and who have received two or more prior therapeutic regimens. There will be no intra-patient dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HL or ALCL.
* Patients must have received two or more prior therapeutic regimens, one of which should include hematopoietic cell transplant, either autologous or allogeneic transplant.
* If a hematopoietic cell transplant was refused, or the patient was not eligible to receive a transplant, the patient is still eligible to participate in the trial if the patient has received two or more prior chemotherapy based regimens.
* Patients who have received allogeneic transplant must not have relapsed less than 6 months after their transplant and they must be at least 200 days post-transplant prior to enrollment, and with no evidence of GVHD
* Patients should have at least one radiographically measurable site of disease of 1.5 cm in the largest dimension.
* Patients must have completed all anti-cancer treatment > 4 weeks prior to enrollment.
* Patients must have completed any palliative corticosteroid therapy (e.g. for management of Type B symptoms) > 2 weeks prior to enrollment.
* Patients must be 18 years of age.
* Required baseline laboratory data:

  * Platelet count 80,000/mm3 (patients must not be platelet transfusion-dependent as evidenced by maintenance of platelet count above 50,000/mm3 in the 28 days prior to enrollment without transfusion)
  * Absolute neutrophil count > 1,500/mm3
  * Creatinine ≤ 1.5 times ULN
  * ALT (SGPT) /AST (SGOT) ≤ 2.5 times upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 times ULN
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.

Exclusion Criteria:

* Patients with known HL or ALCL involvement of either the leptomeningeal or central nervous system.
* Patients requiring treatment with oral or intravenous corticosteroids or other oral or intravenous immunosuppressive agents.
* Patients that have been designated Class III or IV by the New York Heart Association criteria.
* Patients with a history of myocardial infarction or stroke within the last 6 months.
* Patients with active infection are not eligible. This includes patients requiring anti-infective treatment during the 4 week period prior to enrollment. Patients on prophylactic anti-infective agents will be eligible provided they have no signs of active infection.
* Patients who are known to be HIV, Hepatitis B, or Hepatitis C positive.
* Patients with a history of prior malignancy other than HL or ALCL that have not been in remission for greater than 5 years, with the exception of basal or squamous skin carcinoma, cervical carcinoma in situ on biopsy, or localized prostate cancer (Gleason score < 5).
* Patients who are pregnant or breastfeeding.
* Patients with major surgery or radiation therapy within four weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Identification of the maximum tolerated dose and identification of the recommended dose of XmAb®2513 for evaluation in future studies. | 1 year

SECONDARY OUTCOMES:
Safety and tolerability | 1 year
Assessment of immunogenicity | 1 year
Objective response rate, disease control rate, and progression free survival. | 1 year
Change in solCD30 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anas Younes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Rush University Medical Center, Chicago, Illinois
  - Ohio State University, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas